CLINICAL TRIAL: NCT06215508
Title: Prostate Cancer Geriatric Assessment and Technology Evaluation (ProsGATE) Study
Brief Title: Geriatric Assessment and Technology Evaluation in Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB23-1569
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Questionnaires participants fill out at different study visits

SUMMARY:
By doing this study, doctors hope to learn more about factors that contribute to frailty (a condition where older adults feel weak, get tired easily, and struggle more with everyday activities) and serious side effects among men over the age of 65 who will receive androgen deprivation therapy (also called "hormone therapy") for prostate cancer that has spread to other parts of their body. Participation in this research will last about 5 years. For the first year, participants will have 5 study visits where they have give blood samples, answer survey questions, and use a wearable device. After study visits are complete, there is a 4-year follow-up period. Research team will check regular doctor visits and look at participants' medical records.

DETAILED DESCRIPTION:
By doing this study, doctors hope to learn more about factors that contribute to frailty (a condition where older adults feel weak, get tired easily, and struggle more with everyday activities) and serious side effects among men over the age of 65 who will receive androgen deprivation therapy (also called "hormone therapy") for prostate cancer that has spread to other parts of their body. Participation in this research will last about 5 years. For the first year, participants will have 5 study visits where they have give blood samples, answer survey questions, and use a wearable device. After study visits are complete, there is a 4-year follow-up period. Research team will check regular doctor visits and look at participants' medical records.

The purpose of this research is to gather information about the physical, mental, and social health of study participants to help the research team identify factors that put older men with prostate cancer at greater risk for developing serious side effects during hormone therapy. This study is for individuals who are over the age of 65 and plan to receive hormone therapy as part of standard treatment for their prostate cancer. Participants will receive androgen deprivation therapy as part of their standard care with their doctor outside of this study. No drugs or treatments will be given in this study. Participants will instead fill out questionnaires, provide blood samples, and wear a smartwatch paired to a mobile application downloaded to the their personal smartphone or a phone/tablet provided by the research team. This application will help the research team collect information about each study participants' levels of function, general health, physical activity, body composition, memory, mood and side effects during hormone therapy. By collecting this information, doctors leading the study ultimately hope to learn new ways to potentially improve treatment options for older men with prostate cancer while lowering their risks for serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of prostatic origin without neuroendocrine differentiation or signet ring or small-cell histologic features.
* Patients must be metastatic by having at least one metastatic lesion seen at the time of diagnosis or upon initiation of treatment on bone scan or computed tomography (CT) or magnetic resonance imaging (MRI), or by next-generation molecular imaging (FDG, F-18 sodium fluoride (NaF), C-11 choline, F-18 Fluciclovine, Ga-68 Prostate-specific membrane antigen (PSMA-11) positron emission tomography/computed tomography or magnetic resonance imaging.
* Age ≥ 65years. positron emission tomography the aforementioned GA tools are only validated in those aged 65 and older.
* Planned initiation of intensified hormone deprivation (ADT and ARSI)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with previous exposure to ADT/ARSI within 12 months of diagnosis, except those who initiated ADT/ARSI within 12 weeks of enrollment.
* Participants who had surgical orchiectomy outside of 12 weeks before their metastatic diagnosis.
* Participants who have had previous chemotherapy for metastatic prostate cancer.
* Uncontrolled intercurrent illness. "Uncontrolled intercurrent illness" refers to a concurrent medical condition that is not adequately managed or stable at the time of enrollment. This could be any illness, disorder, or medical issue occurring alongside the primary disease being treated or studied, and its lack of control poses additional risk to the patient or complicates the management of the primary condition. For example, in the context of enrolling patients in a clinical trial for a cancer treatment, a patient with uncontrolled diabetes mellitus or hypertension would be considered to have an uncontrolled intercurrent illness as diabetes and hypertension - if poorly managed - can lead complications that could interfere with the patient's ability to safely participate in the trial, potentially confounding the study results or posing additional health risks to the patient.
* Participants with small-cell carcinoma of the prostate or brain metastasis.
* Participants who are not fluent in reading/writing English or Spanish.
* Biologic and Pregnant women are excluded from this study because prostate cancer is a disease of biological males.
* Participants with implantable cardiac devices.
* Participants with limb defects precluding smart-watch wear.

Min Age: 18 Minutes | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: participants with metastatic prostate cancer over the age of 65
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Cancer and Aging Research Group (CARG) scores | 5 years
  To determine if Cancer and Aging Research Group (CARG) scores (≤5 or >5) correlate with vulnerability as classified by comprehensive geriatric assessment (GA) International Society of Geriatric Oncology 2 (SIOG2) criteria, in older participants with metastatic hormone-sensitive prostate cancer (mHSPC) initiating treatment with androgen receptor signaling inhibitors (ARSI).

SECONDARY OUTCOMES:
Serious Adverse Events | 5 years
  To evaluate the relationship between baseline CARG scores in predicting serious adverse events (SAEs) incidence over 12 months in older participants with metastatic hormone-sensitive prostate cancer (mHSPC) patients initiating ARSI therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- o University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF